CLINICAL TRIAL: NCT05393622
Title: Intracalvarial Prefrontal Cortical Stimulation in Treatment-Resistant Depression
Brief Title: Brain Stimulation for Severe Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Inner Cosmos Inc (Industry)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: G210101
Record Dates: First submitted 2022-05-23; First posted 2022-05-26 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2023-10

CONDITIONS: Depression Severe

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Intervention, Placement of Device & Stimulation (Experimental): Placement of neurostimulation device & stimulation of prefrontal cortex target
  Interventions: Device: INTRACALVARIAL PREFRONTAL CORTICAL STIMULATION (IpCS) IN SEVERE TREATMENT-RESISTANT DEPRESSION

INTERVENTIONS:
Device: INTRACALVARIAL PREFRONTAL CORTICAL STIMULATION (IpCS) IN SEVERE TREATMENT-RESISTANT DEPRESSION — Subjects will have the neurostimulation device placed in the skull and continuous stimulation will be applied to relieve symptoms of depression.

SUMMARY:
Chronic intracalvarial cortical stimulation is a minimally invasive method involving the neurosurgical placement of an electrode above the inner table of the skull. Over time, intracalvarial cortical stimulation is intermittently activated to modulate locally and distally connected brain regions. Because of the important role played by the dorsolateral prefrontal cortex in mood regulation, the goal of this study is to apply intracalvarial prefrontal cortical stimulation (IpCS) over the dorsolateral prefrontal cortex in severely treatment-resistant depressed (TRD) patients. Per the DSM-V and Centre for Medicare and Medicaid Services (CMS) nomenclatures, TRD patients are commonly defined as those whose treatment failed to produce response or remission after 2 or more attempts of sufficient duration and treatment dose.

In the investigator's study, eligible TRD subjects will have a diagnosis of major depressive disorder with a suboptimal response to an adequate dose and duration of at least two different antidepressant treatment categories. These subjects will also have had exposure and transiently (non-durably) responded to non-invasive neurostimulation. The investigator anticipates that severely Treatment Resistant Depressed (TRD) Subjects with IpCS of the dorsolateral prefrontal cortex will show a significant decrease in depression symptoms as measured by the Montgomery-Asberg Depression Rating Scale (MADRS) at four months post-implant when compared to baseline.

The investigator will enroll up to 20 subjects with severe refractory depression in an open trial, followed for up to one year. Depressive and cognitive symptoms will be rated periodically to assess the safety and efficacy of this procedure.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for this study, a subject must meet all the following inclusion:

1. Subject has a diagnosis of chronic (≥ two years) or recurrent (multiple prior episodes) depression and is currently experiencing a major depressive episode as defined by DSM V criteria.
2. Subject meets a pre-treatment baseline threshold with MADRS score of >/=20
3. Subject has not had an sustained response to two or more adequately dosed antidepressant treatments from at least two different antidepressant treatment classes in the current depressive episode according to the Antidepressant Treatment History Form (ATHF) (Gaynes, 2020).
4. The subject has completed all baseline testing to determine eligibility for the implant surgery (approximately 3 & 2 weeks prior to expected date for implant surgery, CT & MRI brain scans and cognitive testing).
5. Female subject is not pregnant, agrees to use adequate birth control, or is not capable of becoming pregnant (e.g. post-menopausal, no uterus, ligation of fallopian tubes, surgical removal of ovaries)
6. Subject is between the ages of 21 and 80.
7. Subject is able to complete the evaluations needed for this study including the high resolution CT and MRI brain imaging scans.
8. Subject is able to provide written informed consent and has signed the consent form for participation in this study.

Exclusion Criteria:

The presence of any of the following will exclude a subject from the study:

1. The IpCS would (in the investigator's judgment) pose an unacceptable surgical or medical risk for the patient.
2. Subject is expected to require full body magnetic resonance imaging (MRI) during the clinical study.
3. Subject is judged by the investigator to be acutely suicidal (e.g., within the 30 days prior to the IpCS implant, the subject has made a suicide attempt or gesture or has made specific plans or preparation to commit suicide).
4. Subject has a history of schizophrenia, schizoaffective disorder, or other psychotic disorder, or a current major depressive episode that includes psychotic features (commonly referred to as psychotic depression) according to the DSM V criteria.
5. Subject has a neurological disorder like Epilepsy, Dementia, Delirium, Amnestic disorder, and cognitive impairment.
6. Subject has a history of brain injury that resulted in cognitive impairment.
7. Subject has history of bony disorders (changes in bone density may impact the safe and effective use of the device as well a device implantation).
8. Female subjects with a positive urine pregnancy test.
9. Subject is taking a MAO inhibitor drug e.g., Isocarboxazid (Marplan), Phenelzine (Nardil), Selegiline (Emsam), or Tranylcypromine (Panate) that may pose risk for general anesthesia. The Coordinator will Identify MAOI drug and discuss with PI.
10. Subject and/or Subject's psychiatrist DISAGREES with holding constant the subject's ongoing pharmacotherapy for 4 months following enrollment.
11. Presence of hyperostosis frontalis interna (operationally defined, frontal bone thickening of >20mm), as determined by CT scan of the head, at the proposed site of the electrode implantation

5.3 Prohibited Therapy During Study Period No drug is prohibited, with the exception of Monoamine oxidase inhibitors (MAOIs) if they are posing a risk for general anesthesia. If a subject presents on a MAOI, this will be brought to the PI's attention for discussion with the anesthesiologist. Subjects will follow study protocol of IpCS-D. In brief, after enrolling in the IpCS-D study, all subjects will have their ongoing pharmacotherapy held constant for four months. After the 4 months, all drugs for treating mood disorders are allowed.

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-07-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in depression symptoms | 12 months
  Endpoints for depression will be response and remittance, assessed by Montgomery Asberg Scale for Depression.The minimum and maximum values of the Montgomery Asberg Scale for Depression are ___0___ and ___60__. A higher value means more severe depression.

SECONDARY OUTCOMES:
Change in cognitive function | 12 months
  Endpoints for cognitive remediation will be global cognitive performance, measured by the National Institutes of Health Cognition Battery. The minimum and maximum values of the National Institutes of Health Cognition Battery are __0___ and __40__. A higher value means a better outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Jon Willie, MD, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University in St Louis School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No